CLINICAL TRIAL: NCT01734187
Title: Efficacy and Safety of Fermented Cinnamon Vine Powder on Decrement of Body Fat
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chonbuk National University Hospital (Other)
Responsible Party: Principal Investigator, Soo-Wan Chae, Principal Investigator, Clinical Trial Center for Functional Foods, Chonbuk National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CHEVIGEN-OBESE-DB
Record Dates: First submitted 2012-11-22; First posted 2012-11-27 (Estimated); Last update posted 2019-09-03 (Actual); Status verified 2019-08

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fermented Cinnamon Vine Powder (Experimental)
  Interventions: Dietary Supplement: Fermented Cinnamon Vine Powder
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Fermented Cinnamon Vine Powder — Fermented Cinnamon Vine Powder (30g/day)
  Arms: Fermented Cinnamon Vine Powder
Dietary Supplement: Placebo — Placebo (30g/day)
  Arms: Placebo

SUMMARY:
The investigators performed a 12-week, randomized, double-blind, placebo-controlled human trial to evaluate the efficacy and safety of Fermented Cinnamon Vine Powde on decrement of body fat. The investigators measured decrement of body fat parameters , including abdominal fat, Body Fat Mass, LDL-C, HDL-C, Total Cholesterol and triglyceride, and monitored their blood pressure.

ELIGIBILITY:
Inclusion Criteria:

* Males and females 19-55 years old
* BMI(body mass index) ≥ 25 kg/m^2 or WC(Waist Circumference) ≥ 90(men), WC ≥ 85(women)
* Able to give informed consent

Exclusion Criteria:

* Significant variation in weight(more 10%) in the past 3 months
* Allergic or hypersensitive to any of the ingredients in the test products
* History of reaction to any of the test products or of gastrointestinal diseases such as Crohn's disease or gastrointestinal surgery
* History of alcohol or substance abuse
* Participation in any other clinical trials within past 2 months
* Laboratory test, medical or psychological conditions deemed by the investigators to interfere with successful participation in the study
* Pregnant or lactating women etc.

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2012-01-02 (Actual); Primary Completion 2014-05-29 (Actual); Study Completion 2014-05-29 (Actual)

PRIMARY OUTCOMES:
Changes in abdominal Fat | 12 weeks
  Abdominal Fat was measured in study visit 1(0 week) and visit 3(12 week).
Changes in Body Fat Mass | 12 weeks
  Body Fat Mass was measured in study visit 1(0 week) and visit 3(12 week).

SECONDARY OUTCOMES:
Changes in LDL-cholesterol(Low Density Lipoprotein - Cholesterol) | 12 weeks
  LDL-C(Low Density Lipoprotein - cholesterol) was measured in study visit 1(0 week) and visit 3(12 week).
Changes in HDL-Cholesterol(High Density Lipoprotein - Cholesterol) | 12 weeks
  HDL-cholesterol(High Density Lipoprotein - cholesterol) was measured in study visit 1(0 week) and visit 3(12 week).
Changes in total cholesterol | 12 weeks
  Total cholesterol was measured in study visit 1(0 week) and visit 3(12 week).
Changes in Triglycerides | 12 weeks
  Triglyceride was measured in study visit 1(0 week) and visit 3(12 week).

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Trial Center for Functional Foods; Chonbuk National University Hospital, Jeonju, Jeollabuk-do, South Korea